CLINICAL TRIAL: NCT05711082
Title: MONITORING OF REALITY AND DOPAMINE: A PHARMACOLOGICAL RESEARCH
Brief Title: REALITY MONITORING
Acronym: MORDOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-A01345-38
Record Dates: First submitted 2023-01-23; First posted 2023-02-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Neurosciences

STUDY DESIGN:
Intervention Model Description: MORDOR study will use a randomized, double dummy, placebo-controlled, three-arm crossover design.
Who Masked: Participant
Masking Description: double dummy, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dopamine precursor (Active Comparator): In the first condition, volunteers will receive a dopamine (DA) precursor (L-dopa, 100mg). L-dopa will be combined with a dose of an Aromatic amino acid decarboxylase inhibitor (Benserazide) 25mg to multiplicate its bioavailability and with a dose of domperidone 10mg (peripheral antagonist of DA) to minimize the risk of side effects.
  Interventions: Other: Précurseur de la dopamine
- D2 antagonist (Active Comparator): In the second condition, volunteers will receive a D2 antagonist (Sulpiride, 800mg)
  Interventions: Other: antagoniste D2
- PLACEBO (Placebo Comparator): In the third condition, volunteers will receive a placebo (lactose)
  Interventions: Other: PLACEBO

INTERVENTIONS:
Other: Précurseur de la dopamine — In the first condition, volunteers will receive a 100mg dose of L-dopa, 25mg dose of Aromatic amino acid decarboxylase inhibitors (Benserazide) and 10mg dose of Domperidone. In the second condition, volunteers will receive Sulpiride 800mg. In the third condition, volunteers will receive placebo Reality-monitoring performances will be evaluated with a standardized task. Working-memory will be evaluated with the n-back task. Self-monitoring performances will be observed during a speech production experiment in which speakers monitor their auditory feedback while speaking.
  Speech Bayesian reasoning: This task is a home-made task investigating the influence of prior on speech processing. Subjects will be required to identify speech in ambiguous auditory stimuli. Visual Bayesian reasoning: This task investigates the influence of prior on visual processing. Subjects will be required to recognize morph between faces and house.
  Arms: Dopamine precursor
Other: antagoniste D2 — In the second condition, volunteers will receive Sulpiride 800 mg
  Arms: D2 antagonist
Other: PLACEBO — In the third condition, volunteers will receive placebo
  Arms: PLACEBO

SUMMARY:
Reality-monitoring characterizes the ability to determine whether information was perceived in the environment or only imagined . Impaired reality-monitoring abilities have been associated with hallucinations in patients with schizophrenia and patients with Parkinson's disease.

The investigators hypothesize a link between dopaminergic (DA) transmission and reality-monitoring.

DETAILED DESCRIPTION:
This hypothesis is based on several studies in the literature: 1) DA transmission anomalies are observed in both schizophrenia and Parkinson's disease; 2) DA agonists may induce hallucination; 3) DA antagonists reduce hallucinations and improve reality-monitoring abilities in patients with schizophrenia. In addition, also suggesting a link between mesocorticolimbic connectivity, subcortical DA transmission and reality-monitoring, The investigators have shown that fronto-temporal transcranial Direct Current Stimulation (tDCS) leads:

* on the one hand, to modulate reality-monitoring performance in healthy volunteers and patients;
* on the other hand, to induce subcortical DA release. However, to date, no study has yet explored the direct link between DA transmission and reality-monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who have given their written informed consent
* Men and women from 18 to 45 years old
* Normal or corrected vision
* Being fluent in French or French for native language
* Being affiliated with health insurance

Exclusion Criteria:

* Healthy volunteers who have given their written informed consent
* Men and women from 18 to 45 years old
* Normal or corrected vision
* Being fluent in French or French for native language
* Being affiliated with health insurance
* Inadmissibility of the subject's consent or refusal
* Working-memory deficit (as controlled with MMSE score< 23)
* Any past or current psychiatric or somatic condition(as controlled with the Mini International Neuropsychiatric Interview, MINI)
* Any past or current neurological condition
* History of cranio-cerebral trauma, arterial hypotension or hypertension, cardiological or serious medical condition
* Abnormal potassium dosage (below 3.1 mmol/L or above 4.9 mmol/L)
* Anormal ECG
* History of schizophrenia or bipolar disorder in first-degree relatives
* Alcohol-drinking and caffeine intake at least during 24 hours before each session
* Drug therapy excepting contraceptives
* Cardiologic or severe medical conditio
* Pregnancy(checked with a pregnancy autotest), lactation, or insufficient contraceptive measure (precautionary measure)
* Consumption of recreational drugs during the last 6 months
* Known sensitivity to any of the study medication and their excipients
* Lactose intolerance
* Porphyria
* Hepatic insufficiency

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reality-monitoring performance | One month
  Measured with a behavioral task developed, validated and used in investigators lab.
  During the memory retrieval phase, 48 words will be presented, including the 32 words presented during encoding as well as 16 new words. Subjects will be required to identify whether each word was previously heard, imagined or new. Three words lists will be used and assigned randomly depending on the substance condition (L-dopa, Sulpiride, placebo). Each verbal list will include 16 items with the "imagine hear" encoding condition and 16 items with the "listen" encoding condition.
  A single measure including two variables of interest will account for the main evaluation criteria:
  * The average conditional source-identification measure (ACSIM) which represents the overall ability to correctly retrieve the source, conditional on that item was recognized as already presented.
  * The source misattributions,the number of confusions between heard and imagined events.

SECONDARY OUTCOMES:
Reaction times at the reality-monitoring task and scores of subjective confidence rating for reality-monitoring responses | One month
  Regarding reality-monitoring, a single test in which investigators will also measure the reaction times at the reality-monitoring task and scores of subjective confidence rating for reality-monitoring responses. The variable of interest will be the number of high-confident incorrect source-recognition responses. Investigators finally measure the vividness of each "imagined" or "listened" word with Visual Analogue Scales (VAS) from 0 to 100.
Other cognitive tasks | One month
  In the same test investigators will measure the number of correct/incorrect responses and reaction times at the n-back working memory task.
  * The effect of dopamine modulation on the ability the ability to determine our speech as self-generated will be measured with a self-monitoring task. Investigators measure the magnitude of a voice peak response reflecting the feeling of agency.
  * The effect of dopamine modulation on perception will be evaluated with the performances measured during 2 home-made Bayesian reasoning tasks, evaluating speech processing and visual processing, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: FILIPE GALVAO, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No